CLINICAL TRIAL: NCT01409928
Title: A Study of the Laparoscopically-placed Adjustable Gastric Band for the Management of Obesity in Adolescent Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 102010-093
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Obesity
Keywords: obesity; adolescent; pediatric; weight loss; bariatric surgery; gastric banding
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lap-Band (Experimental): Placement of the LAP-BAND® system will be performed laparoscopically under general anesthesia, using the pars flaccida technique. The device will be placed by surgeons from the University of Texas Southwestern Medical Center Obesity Management Program at Children's Medical Center Dallas. Surgeons will be fully trained in the placement of the LAP-BAND® device, in accordance with FDA approval of the device for the placement in adults. As is current practice in adults undergoing the procedure, incidentally discovered hiatal hernias are repaired at the time of band placement, to reduce the incidence of post-operative reflux. Children receive prophylactic antibiotics, and are observed overnight after surgery. Patients are generally discharged from the hospital the next day. The band will initially be left empty at the end of the placement procedure.
  Interventions: Device: LAP-BAND (Allergan, Inc.)

INTERVENTIONS:
Device: LAP-BAND (Allergan, Inc.) — Laparoscopic placement of adjustable gastric banding system for the treatment of severe obesity.
  Other Names: Lap-Band Adjustable Gastric Banding System

SUMMARY:
This is a prospective, non-randomized, single center study of a laparoscopically placed, adjustable gastric band medical device for the treatment of adolescent obesity.

DETAILED DESCRIPTION:
Study population We plan to enroll 30 subjects between the ages of 14 and 17 years with the LAP-BAND®. The inclusion criteria are in accordance with recent evidence-based indications for the surgical management of severe obesity in the pediatric population (Pratt, Lenders et al. 2009). The enrollees will be children who have a body-mass index in the 99th percentile, corresponding to a BMI>= 35 kg/m2, and who exhibit significant comorbidities.

This sample size will provide over 90% power to detect a 15% change in body mass index with a standard deviation of 6, two-tailed alpha of 0.05, and allow for 20% loss to follow-up, using a paired design.

ELIGIBILITY:
Inclusion Criteria:

* BMI >= 35 kg/m2 and at least one serious comorbidity (type 2 diabetes mellitus, moderate or severe obstructive sleep apnea, pseudotumor cerebri, and severe steatohepatitis)
* BMI => 40 kg/m2 and a serious comorbidity (as listed above or at least one other comorbidity (mild obstructive sleep apnea, hypertension, insulin resistance, glucose intolerance, dyslipidemia, impaired quality of life or activities of daily living)
* Must live in Dallas/Fort Worth area so that necessary follow-up can be ensured.

Exclusion Criteria:

* Intention to have another surgical procedure for weight reduction within 12 months of LAP-BAND® placement
* History of pregnancy, or the intention to become pregnant within the next 12 months
* History of substance abuse within one year prior to surgery
* Obesity caused by medically correctable condition
* History of gastric or esophageal surgery, or the presence of an esophageal dysmotility disorder
* Eating disorder that is untreated
* Chronic use of aspirin and/or nonsteroidal anti-inflammatory medications and unwillingness to discontinue the use of these medications
* History of previous bariatric surgery, intestinal obstruction, or peritonitis
* Presence of localized or systemic infection at the time of surgery
* History of congenital or acquired anomalies of the gastrointestinal tract
* History of immunocompromise, or auto-immune, hematologic or dermatologic condition that increases risk of bleeding, breakdown of skin integrity (due to port), or infection.
* Planning to or having high likelihood of moving out of region within 2 years
* Portal Hypertension or Cirrhosis
* Uncorrectable coagulopathy or severe bleeding disorder
* Use of weight loss medications within 6 weeks of procedure

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-03-21 (Actual); Study Completion 2016-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perrin White, Principal Investigator — UTSW
Locations (1):
- Children's Medical Center Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lap-Band
Started | 16
Completed | 4
Not Completed | 12
Not completed — Physician Decision | 12

BASELINE CHARACTERISTICS:
Arm/Group | Lap-Band
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index Z-score
Description: Measure of relative weight adjusted for child age and sex. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: 12 months post operation
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Lap-Band
Number analyzed (Participants) | 4
Z-score | -0.26 (0.21)

ADVERSE EVENTS:
Arm/Group | Lap-Band
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No